CLINICAL TRIAL: NCT00989586
Title: A Phase I/II Study of Veltuzumab (IMMU-106, hA20), a Humanized Anti-CD20 Monoclonal Antibody, Combined With Milatuzumab (IMMU-115, hLL1), a Humanized Anti-CD74 Monoclonal Antibody, in Relapsed and Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Veltuzumab and Milatuzumab in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Christian (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Beth Christian, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09024; NCI-2011-03150 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; MALT lymphoma; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; Waldenstrom macroglobulinemia
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — milatuzumab; Antibodies, Monoclonal; veltuzumab; Blood Specimen Collection; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental): Phase I portion of the study, a standard 3+3 dose escalation schema will be followed. Patients will receive veltuzumab IV weekly on day 1 for 4 doses and milatuzumab weekly on for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive veltuzumab alone on day 1 and milatuzumab alone on day 2 to prevent overlapping infusion reactions. Starting week 2, veltuzumab will be given on day 1 and milatuzumab will be given on day 4.
  Interventions: Biological: milatuzumab; Biological: veltuzumab; Procedure: Correlative/Special Studies; Procedure: Quantitative T-, B-, and NK cell subsets; Procedure: Pharmacokinetics; Procedure: Human Anti-Human Antibodies
- Phase II (Experimental): Patients will receive veltuzumab IV weekly for 4 doses and milatuzumab IV weekly on day 2 of week 1 and on day 4 of weeks 2-4 for 4 total doses during induction therapy. Patients may continue on therapy to receive extended induction therapy provided they do not experience significant toxicity or rapid disease progression during the initial 4 week induction.
  Interventions: Biological: veltuzumab and milatuzumab

INTERVENTIONS:
Biological: milatuzumab — Patient will receive milatuzumab weekly for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive milatuzumab on day 2. Starting in week 2, milatuzumab will be given on day 4. Provided the patient does not experience excessive toxicity or disease progression during induction therapy, the patient may continue treatment with extended induction therapy, consisting of veltuzumab day 1 and milatuzumab day 4 of weeks 12, 20, 28, and 36.
  Other Names: monoclonal antibody
  Arms: Phase I
Biological: veltuzumab — Patient will receive veltuzumab weekly for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. Provided the patient does not experience excessive toxicity or disease progression during induction therapy, the patient may continue treatment with extended induction therapy, consisting of veltuzumab day 1 and milatuzumab day 4 of weeks 12, 20, 28, and 36.
  Other Names: monoclonal antibody
  Arms: Phase I
Procedure: Correlative/Special Studies — To correlate Fcγ receptor polymorphisms with response to treatment with the combination of veltuzumab and milatuzumab. Whole blood will be collected pre-treatment on day 1.
  Other Names: blood samples
  Arms: Phase I
Procedure: Quantitative T-, B-, and NK cell subsets — Quantitative T-, B-, and NK- cell subsets will be assessed using flow cytometry to quantify the percentage and absolute number of cells expressing CD4, CD8, CD56, CD16, CD19, and CD20 pre-treatment on day 1, after induction (week 5, day 1), and prior to the start of therapy on day 1 week 12, day 1 week 36, and then every 4 months for one year.
  Other Names: blood samples
  Arms: Phase I
Procedure: Pharmacokinetics — To assess the pharmacokinetics of veltuzumab in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma. Pharmacokinetics will be assessed with blood samples collected at the following time points: immediately pre- and post-infusion on day 1 of weeks 1, 2, 4, 12 and 36. One additional sample will be collected each of weeks 5 through 10 (sample may be collected any day during each of these weeks).
  Other Names: blood samples
  Arms: Phase I
Procedure: Pharmacokinetics — To assess the pharmacokinetics of milatuzumab in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma. Pharmacokinetics will be assessed with blood samples collected at the following time points: immediately pre- and post-infusion on day 2 of week 1 and day 1 of weeks 2, 4, 12 and 36. Additional samples will be collected days 3 through 6 of week 1.
  Other Names: blood samples
  Arms: Phase I
Procedure: Human Anti-Human Antibodies — To monitor for the development of human anti-veltuzumab antibodies and human anti-milatuzumab antibodies (HAHA) in patients receiving treatment with veltuzumab and milatuzumab. Patients will be monitored for the development of HAHA at the following timepoints: pre-treatment on day 1 of week 1, pre-treatment on day 1 of week 4, pre-treatment on day 1 of week 12, and pre-treatment on day 1 of week 36.
  Other Names: blood samples
  Arms: Phase I
Biological: veltuzumab and milatuzumab — Patient will receive veltuzumab and milatuzumab weekly for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive veltuzumab on day 1 and milatuzumab on day 2. Starting in week 2, veltuxumab will be given on day 1 and milatuzumab will be given on day 4. Provided the patient does not experience excessive toxicity or disease progression during induction therapy, the patient may continue treatment with extended induction therapy, consisting of veltuzumab day 1 and milatuzumab day 4 of weeks 12, 20, 28, and 36.
  Other Names: monoclonal antibody
  Arms: Phase II

SUMMARY:
A phase I dose escalation study of veltuzumab and milatuzumab in relapsed and refractory B-cell NHL. The phase I study will be followed by a pilot phase II study.

DETAILED DESCRIPTION:
A phase I/II study of veltuzumab combined with milatuzumab in relapsed and refractory non-Hodgkin's lymphoma. Both agents are well-tolerated in early phase clinical testing with infusion reactions as the primary observed toxicity. Preclinical testing in vitro and in vivo have demonstrated single agent activity for both veltuzumab and milatuzumab. In mantle cell lymphoma cell lines and SCID mouse models, synergist effects were observed when milatuzumab was combined with rituximab. Veltuzumab has several advantages over rituximab including slower off-rates, shorter infusion times, higher potency, and improved therapeutic responses in animal models. Previous and ongoing clinical investigations support the concept of combining monoclonal antibodies in NHL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell non-Hodgkin lymphoma (NHL), including any of the following:

  * Marginal zone lymphoma
  * Waldenstrom macroglobulinemia (lymphoplasmacytic lymphoma)
  * Follicular lymphoma
  * Mantle cell lymphoma
* Relapsed or refractory disease after ≥ 1 prior therapy
* Patients with rituximab-refractory disease (defined as having less than a partial response to the prior rituximab-containing regimen) or rituximab-sensitive disease (defined as having a complete response or partial response to the last rituximab-containing regimen [provided it has been ≥ 3 months since the last dose of rituximab]) are eligible.
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG)performance status 0-2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1000/μL
  * Platelets ≥ 75,000/μL
  * Total bilirubin ≤ 2.0 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine ≤ 2.0 mg/dL
* Patients who have relapsed after stem cell transplant are eligible for this trial.
* Patients with active Hepatitis B infection are not eligible.
* Non-pregnant and non-nursing. Women of child bearing potential and men must agree to use contraception prior to study entry and for duration of study participation.
* Must possess the ability to understand and the willingness to sign a written informed consent document.

Phase II

-Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension >10 mm or in the case of Waldenstrom's macroglobulinemia, the presence of an IgM paraprotein level 2x the upper limit of normal.

Exclusion Criteria:

* Must be recovered from all toxicities from prior therapy or radiation (excluding alopecia).
* No known CNS lymphoma.
* History of documented human anti-globulin antibodies.
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations.
* HIV-positive patients.
* Pregnant women.
* Patients with secondary malignancies with exception of non-melanomatous skin cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Christian, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christian BA, Poi M, Jones JA, Porcu P, Maddocks K, Flynn JM, Benson DM Jr, Phelps MA, Wei L, Byrd JC, Wegener WA, Goldenberg DM, Baiocchi RA, Blum KA. The combination of milatuzumab, a humanized anti-CD74 antibody, and veltuzumab, a humanized anti-CD20 antibody, demonstrates activity in patients with relapsed and refractory B-cell non-Hodgkin lymphoma. Br J Haematol. 2015 Jun;169(5):701-10. doi: 10.1111/bjh.13354. Epub 2015 Apr 7. PMID 25847298
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Phase I portion of the study, a standard 3+3 dose escalation schema will be followed. Patients will receive veltuzumab IV weekly on day 1 for 4 doses and milatuzumab weekly on for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive veltuzumab alone on day 1 and milatuzumab alone on day 2 to prevent overlapping infusion reactions. Starting week 2, veltuzumab will be given on day 1 and milatuzumab will be given on day 4.
  milatuzumab: Patient will receive milatuzumab weekly for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive milatuzumab on day 2. Starting in week 2, milatuzumab will be given on day 4. Provided the patient does not experience excessive toxicity or disease progression during induction therapy, the patient may continue treatment with
- Phase II: Patients will receive veltuzumab IV weekly for 4 doses and milatuzumab IV weekly on day 2 of week 1 and on day 4 of weeks 2-4 for 4 total doses during induction therapy. Patients may continue on therapy to receive extended induction therapy provided they do not experience significant toxicity or rapid disease progression during the initial 4 week induction.
  veltuzumab and milatuzumab: Patient will receive veltuzumab and milatuzumab weekly for 4 total doses during induction therapy. Induction therapy will be defined as the first 4 weeks of study therapy. During week 1 of induction therapy, patients will receive veltuzumab on day 1 and milatuzumab on day 2. Starting in week 2, veltuxumab will be given on day 1 and milatuzumab will be given on day 4. Provided the patient does not experience excessive toxicity or disease progression during induction therapy, the patient may continue treatment with extended induction therapy, consisting of veltuzumab day 1 and milatuzumab day 4 of weeks
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with histologically confirmed B-cell NHL including marginal zone lymphoma, Waldenstrom's macroglobulinemia or lymphoplasmacytic lymphoma, follicular lymphoma, or mantle cell lymphoma by WHO criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 81] | 63 [39 to 82] | 63 [39 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: patients]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) for Phase I Patients
Description: Dose-limiting toxicity was assessed during induction therapy for phase I.
Time Frame: up to 2 years
Measure: Number; unit: patients
Arm/Group | Phase I
Number analyzed (Participants) | 18
patients | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)for Phase I Patients
Description: Patients received a fixed dose of Veltuzumab IV 200 mg/m2 and Milatuzumab was dose escalated
Time Frame: up to 2 years
Measure: Number; unit: mg/kg
Arm/Group | Phase I
Number analyzed (Participants) | 18
mg/kg | 20

3. Primary Outcome: Overall Objective Response Rate
Description: Per International Response Criteria (Cheson JCO 2007) for target lesions and assessed by CT, MRI or PET: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Number; unit: percent of patients
Groups:
- All Patients From Phase I and Phase II: Phase I: patients receive Veltuzumab IV weekly on day 1 for 4 doses and Milatuzumab weekly for total of 4 doses during induction therapy. Induction therapy during week 1 patients receive Veltuzumab alone on day 1 and Milatuzumab alone on day 2 to prevent overlapping infusion reactions. Week 2 Veltuzumab on day 1 and Milatuzumab on day 4.
  Phase II: patients receive Veltuzumab IV weekly for 4 doses and Milatuzumab IV weekly on day 2 of week 1 and on day 4 of weeks 2-4 for 4 total doses during induction therapy.
Arm/Group | All Patients From Phase I and Phase II
Number analyzed (Participants) | 34
percent of patients | 24

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using International Response Criteria (Cheson JCO 2007), as a >= 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or at least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis, or the size of other lesions (eg, splenic or hepatic nodules), or the appearance of new lesions.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients From Phase I and Phase II
Number analyzed (Participants) | 34
months | 4.7 [2.2 to 9.3]

5. Secondary Outcome: Fcγ-receptor Polymorphism Response to Treatment
Description: The relationship between overall response rate (ORR) and Fcy receptor status. A two-sided chi-square test or exact test with α = 0.05 will be used to test the homogeneity of the ORR among the three genotypes.
Time Frame: up to 2 years
Population: This data is not available due to analysis was not performed. The response rate was to low for the analysis to yield results to report for this trial.
Arm/Group | All Patients From Phase I and Phase II
Number analyzed (Participants) | 0

6. Secondary Outcome: Quantitative T-, B-, and NK-cell Subsets Using Flow Cytometry
Description: Quantitative T-, B-, and NK- cell subsets will be assessed using flow cytometry to quantify the percentage and absolute number of cells expressing CD4, CD8, CD56, CD16, CD19, and CD20 at screening, after induction, and prior to the start of therapy on day 1 week 12, day 1 week 28, and then every 4 months for one year.
Time Frame: up to 1 year
Population: as for outcome 5
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Access Pharmacokinetics Through AUC0-∞ (Area Under Curve)
Description: Evaluation of pharmacokinetics (Pk) of veltuzumab and milatuzumab was performed for patients included in the trial. Statistically, descriptive data of PK parameters will be computed. Relationships between such parameters as dose and AUC, volume of distribution, clearance, and others will be evaluated, but be preliminary due to the small sample size.
Time Frame: 0, 24, 48, 72, 96 and 120 hours post-does
Population: AUC0-∞ for patients dosed at 20 mg/kg
Measure: Mean (Standard Deviation); unit: d*ug/ml
Groups:
- Patients Dosed at 20mg/kg: First dose milatuzumab pharmacokinetics for patients doses at 20 mg/kg
Arm/Group | Patients Dosed at 20mg/kg
Number analyzed (Participants) | 17
d*ug/ml | 422 (121)

8. Secondary Outcome: Access Pharmacokinetics Through Cmax
Description: Evaluation of pharmacokinetics of veltuzumab and milatuzumab was performed for patients included in the trial. Statistically, descriptive data of PK parameters will be computed. Relationships between such parameters as dose and AUC, volume of distribution, clearance, and others will be evaluated, but be preliminary due to the small sample size.
Time Frame: 0, 24, 48, 72, 96 and 120 hours post-dose
Population: Cmax for patients dosed at 20 mg/kg
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Patients Dosed at 20mg/kg
Number analyzed (Participants) | 17
ug/ml | 480 (116)

9. Secondary Outcome: Monitor Human Anti-veltuzumab Antibodies and Human Anti-milatuzumab (HAHA)
Description: Patients will be monitored for the development of human anti-veltuzumab antibodies and human anti-milatuzumab antibodies (HAHA).
Time Frame: up to 36 weeks
Population: HAHA titres were assayed for patients in Phase I and Phase II
Measure: Number; unit: patients
Arm/Group | All Patients From Phase I and Phase II
Number analyzed (Participants) | 33
patients
  anti-veltuzumab antibodies | 1
  anti-milatuzumab antibodies | 0

ADVERSE EVENTS:
Description: Adverse event grading was done according to NCI CTCAE version 3.0 as classified either possibly, probably, or definitely related to study treatment.
Groups:
- All Patients From Phase I and Phase II: Toxicities were graded according to NCI Common Toxicity Criteria for Adverse Events version 3.0 and classified as either unrelated, unlikely, possibly, probably or definitely related to study treatment.
Arm/Group | All Patients From Phase I and Phase II
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients From Phase I and Phase II (N=35)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion Reaction (Injury, poisoning and procedural complications) | 3 (3)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Death (General disorders) | 2 (2) — due to disease progression within 30 days of treatment
Fatigue (General disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Fever without neutropenia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients From Phase I and Phase II (N=35)
Leukopenia (Blood and lymphatic system disorders) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 19 (19)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7)
Infection (Infections and infestations) | 5 (5)
Infusion Reactions (Injury, poisoning and procedural complications) | 21 (21)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Chills (General disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes